CLINICAL TRIAL: NCT04141787
Title: Ceftriaxone as Home Intravenous Therapy for Deep-Seated Staphylococcal Infections, a Randomized Non-Inferiority Trial
Brief Title: Ceftriaxone as Home IV for Staph Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Eric Partlow, Infectious Diseases Physician (Section Chief), Vancouver Island Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C2018-018
Record Dates: First submitted 2019-10-17; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Staphylococcal Infections; Osteomyelitis; CNS Infection; Septic Arthritis; Diabetic Foot Infection; Vertebral Osteomyelitis; Abscess; Coagulase Negative Staphylococcal Infection
Keywords: Ceftriaxone; Deep-seated Infections; Staphylococcus aureus; Coagulase-negative Staphylococcus species; MSSA; CoNS
MeSH Terms: conditions — Staphylococcal Infections; Osteomyelitis; Central Nervous System Infections; Arthritis, Infectious; Abscess | interventions — Ceftriaxone; Cloxacillin; Cefazolin; Daptomycin

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, unblinded non-inferiority trial being led by infectious diseases clinicians. We have chosen a pragmatic trial design which represents the most efficient use of available resources to test the study hypothesis and is the designed to determine effectiveness as opposed to efficacy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftriaxone (Active Comparator): Ceftriaxone 2g IV q24hvia Gravity (or q12h in the case of CNS infections) Duration dependent on site of infection, determined by treating infectious diseases (ID) clinicians based on accepted clinical guidelines.
  Interventions: Drug: Ceftriaxone
- Usual Antibiotics (Cloxacillin, Cefazolin, Daptomycin) (Active Comparator): "Usual Antibiotics" to treat methicillin-susceptible Staphylococcal infections
  * Cloxacillin 2g IV q4h via Pump (dose adjusted for renal function)
  * Cefazolin 2g IV q8h via Preloaded Syringe (dose adjusted for renal function)
  * Daptomycin 6-10mg/kg IV daily via Gravity (dose will be determined based on the severity of infection as per discretion of the ID clinician and in accordance with most recent evidence)
  * Duration dependent on site of infection, determined by treating infectious diseases clinicians based on accepted clinical guidelines.
  Interventions: Drug: Usual Antibiotics (Cloxacillin, Cefazolin, Daptomycin)

INTERVENTIONS:
Drug: Ceftriaxone — Participants with methicillin-sensitive deep-seated staphylococcal infections eligible for treatment on home IV will be randomly assigned to a "treatment" group of ceftriaxone or "standard therapy/usual antibiotics" with either cloxacillin, cefazolin or daptomycin. The treatment with one of the three "standard therapies/usual antibiotics" will be left to the discretion of the treating Infectious Disease doctor, in line with current standards of practice.
  Other Names: Rocephin
  Arms: Ceftriaxone
Drug: Usual Antibiotics (Cloxacillin, Cefazolin, Daptomycin) — Participants with methicillin-sensitive deep-seated staphylococcal infections eligible for treatment on home IV will be randomly assigned to a "treatment" group of ceftriaxone or "standard therapy/usual antibiotics" with either cloxacillin, cefazolin or daptomycin. The treatment with one of the three "standard therapies/usual antibiotics" will be left to the discretion of the treating Infectious Disease doctor, in line with current standards of practice.
  Other Names: Cloxacillin; Cefazolin; Daptomycin; Ancef; Cubicin
  Arms: Usual Antibiotics (Cloxacillin, Cefazolin, Daptomycin)

SUMMARY:
Patients who are admitted to hospital with serious infections, such as those in bone, joints or spine, require a long course of intravenous (IV) antibiotics. After an initial treatment course in hospital or through a dedicated outpatient antibiotic program many patients can complete their treatment course at home. Such infections are often caused by bacteria called Staphylococci, and currently there are three antibiotic options used routinely. A fourth antibiotic, ceftriaxone, is a promising alternative; it is also effective against Staphylococci, and is more convenient, less costly and easier to give at home, however, it has not been studied thoroughly in a prospective manner. This study will compare ceftriaxone to routinely used antibiotics (cloxacillin, cefazolin or daptomycin) to see if ceftriaxone is equally as safe and efficacious in curing deep-seated Staphylococcal infections in patients receiving home IV antibiotics. Patients with deep-seated infections caused by methicillin-susceptible Staphylococcus aureus (MSSA) or coagulase-negative Staphylococcal species will be randomly assigned home IV treatment with ceftriaxone OR one of the three other antibiotics before leaving the hospital. Patients will then receive usual care from an Infectious Disease physician and Home IV team. The study team will assess whether cure has been achieved by the end of the IV treatment, follow-up at 6 months to see if patients remain infection-free, and record any side-effects of treatment. The overall goal is to determine whether ceftriaxone can be considered non-inferior to usual antibiotic treatment in treating Staphylococcal infections in a home IV setting.

DETAILED DESCRIPTION:
The use of ceftriaxone for deep-seated Staphylococcal infections requiring prolonged IV treatment is a practice that has already evolved both locally and globally despite the absence of high-quality clinical data. Retrospective studies that support the use of ceftriaxone for this indication, including those that currently inform Infectious Diseases Society of America (IDSA) guidelines, unanimously agree that prospective, randomized data is urgently needed. Our study is the next natural step in the research process and would greatly add to the body of evidence informing this practice by addressing current knowledge gaps. On a clinical level, demonstrating non-inferiority of ceftriaxone would allow its use in a population of patients currently ineligible for outpatient antibiotic treatment or in cases where broader, more expensive agents are currently employed. This would facilitate more rapid discharge from hospital, lead to substantial cost savings, and have a considerable impact on antimicrobial stewardship. Most importantly, it would improve the quality of life of patients by allowing them to be treated at home in cases when multi-dose home IV administration is a barrier to discharge. This study would address the need to support and harmonize current practice at Island Health, increase the level of evidence in current guidelines and improve patient care both locally and globally.

This is a prospective, randomized, controlled, unblinded trial with a pragmatic design. The goal is to assess whether the intervention is non-inferior to standard therapies in achieving the primary outcome. Patients will be drawn from inpatient populations and patients treated through an outpatient antibiotic therapy clinic who are eligible for further IV treatment through a home intravenous therapy program. Patients meeting inclusion criteria as described will be asked to participate and informed consent obtained. Once informed consent is obtained patients will be randomized to receive ceftriaxone or standard therapies (cloxacillin, cefazolin, daptomycin) as determined by the treating infectious diseases physician. Patients will have deep-seated infections such as:

* Osteomyelitis
* Native Joint Septic Arthritis
* Prosthetic Joint Septic Arthritis
* Central Nervous System Infection
* Deep Tissue Infection
* Diabetic Foot Infection

Infections will be confirmed to have been caused by methicillin-sensitive Staphylococcus aureus or a coagulase-negative Staphylococcal species through microbiological testing. Susceptibility testing will ensure that the isolate is susceptible to the study drug and at least one of the standard therapies.

Once the patient is randomized all other aspects of care will follow usual home IV therapy policies and procedures. Neither the patient nor the clinical team will be blinded to the study drug the patient is receiving. Duration of treatment will be decided by the treating infectious diseases clinician based on infection site and available guidelines. Baseline data will be collected by the study team at the time of randomization.

The patient will be followed up in the usual manner by their infectious diseases physician. Data will be collected in a standardized manner at the pre-specified end of antibiotic therapy. Clinical cure (primary outcome) will be determined based on this data.

Adverse event rates will be collected throughout the study period. At six months post-randomization the study team will assess for any markers of treatment failure (see secondary outcomes).

Plan for statistical analysis is pre-specified in the protocol and will be completed with the assistance of biostatistics staff at the University of Victoria. Specific information on the protection of patient confidentiality and data integrity is outlined in the study protocol. Ethics approval has been granted by the Clinical Research Ethics Board at Vancouver Island Health Authority.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older
* were referred to and assessed by an Infectious Disease physician in the form of a clinical consult as either:

  * an inpatient at the Royal Jubilee or Victoria General Hospitals
  * an outpatient at the emergency department of one of the aforementioned hospitals
  * an outpatient at the Outpatient Parenteral Antibiotic Therapy (OPAT) clinic
* have a clinically and/or radiographically diagnosed deep-seated MSSA or coagulase-negative Staphylococcal infection as defined in Table 1 of the protocol (Osteomyelitis, Discitis/Epidural abscess, Central Nervous System (CNS) infection, Abscess, Septic Arthritis (including Prosthetic Joint Infection), Diabetic foot infection) and the diagnosis has been made or confirmed by the Infectious Disease physician
* have had the causative pathogen confirmed microbiologically as either MSSA or CoNS through a laboratory sample indicative of the current site of infection
* are deemed to require prolonged IV antibiotic therapy and subsequently referred for assessment by the home IV program by the Infectious Disease physician
* are an appropriate candidate for the home IV program as determined by the assessing Home IV nurse, and are eligible for treatment with BOTH ceftriaxone AND at least one of the usual alternatives, namely cloxacillin, cefazolin or daptomycin
* provide written informed consent to participate in the study
* have their culture and sensitivity results finalized prior to randomization, with the isolate confirmed to be sensitive to all study drugs (susceptibilities are discussed in the "Microbiological Testing" section of the protocol)
* are successfully randomized to either ceftriaxone OR one of cloxacillin, cefazolin or daptomycin before Home IV orders are written (the choice between the three comparator antibiotics will be at the discretion of the treating Infectious Disease physician)
* receive at least one dose of the antibiotic to which they were randomized prior to being discharged on the home IV program
* are physically discharged to the home IV program for any duration

Exclusion Criteria:

* younger than 18 years of age
* pregnant
* involved in another therapeutic trial
* are not under the care of an Infectious Disease physician
* are unable to provide informed consent due to language or cognitive barriers
* are not appropriate for Home IV therapy as determined by the assessing Home IV nurse
* are concurrently receiving other anti-staphylococcal antibiotics (excluding the synergistic use of rifampin for prosthetic joint infections) at the time of discharge on the home IV program
* have relevant cultures indicating a polymicrobial infection (except in the case of diabetic foot infections where they may be included if MSSA or CoNS is determined to be the dominant pathogen by the Infectious Disease physician and any additional antibiotics used do not exhibit activity against MSSA or CoNS)
* have concurrent or incompletely treated bacteremia with MSSA or CoNS (as defined in protocol)
* have infective endocarditis based on imaging or clinical judgement
* are receiving home IV antibiotics solely as palliative therapy
* are unable to tolerate ceftriaxone AND any ONE of the standardly used antibiotics (cloxacillin, cefazolin, daptomycin) because of an allergy or intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate of deep-seated methicillin sensitive Staphylococcal infections | Up to 6 months post-randomization
  Clinical cure of deep-seated MSSA and CoNS infections will be defined by improvement in clinical parameters, imaging findings and laboratory values at the time of completion of a pre-specified duration of antibiotic treatment based on infection site and clinical guidelines. Clinical cure defined by treating infectious diseases clinicians based on composite of:
  * Resolution of signs and symptoms of deep-seated infection
  * Improvement in inflammatory markers; defined as a C-reactive protein (CRP) less than 50% of initial CRP value
  * Improvement in follow- up imaging when conducted, as determined by the interpreting radiologist

SECONDARY OUTCOMES:
Treatment failure at six months post-randomization | At six months following randomization
  Failure of treatment at six months post-randomization will be defined by:
  * Readmission to hospital for complications or progression of the specific infection being treated
  * Need for further surgical source control procedures
  * Additional antibiotics required for recurrent infection by the same organism, in the same location after initial treatment course was completed
  This will be determined by chart review completed by study team members.
Adverse event rate | Up to 6 months post-randomization
  All adverse events related to study drug with specific safety data on rates of anaphylaxis, Clostridium difficile infections, dermatologic eruptions, hepatic enzyme abnormalities, leukopenia, thrombocytopenia, gastrointestinal upset and acute kidney injury between the two treatment arms.

OTHER OUTCOMES:
Rate of antibiotic substitution or discontinuation | Up to 6 months post-randomization
  If antibiotic needs to be substituted or discontinued for any reason
Duration of therapy | Up to 6 months post-randomization
  Duration of therapy as compared by infection type across both arms

CONTACTS AND LOCATIONS:
Overall Officials: Eric Partlow, MD, FRCPC, Principal Investigator — Vancouver Island Health Authority
Locations (2):
- Canada (2):
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for all primary and secondary outcome measures will be made available within 6 months of study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 months following study completion.
Access Criteria: Access requests will be assessed by a review panel associated with Vancouver Island Health Authority.

REFERENCES:
- [Background] Lother SA, Press N. Once-Daily Treatments for Methicillin-Susceptible Staphylococcus aureus Bacteremia: Are They Good Enough? Curr Infect Dis Rep. 2017 Sep 23;19(11):43. doi: 10.1007/s11908-017-0599-0. PMID 28942574
- [Background] Hotchkies L, Grima DT, Hedayati S. The total process cost of parenteral antibiotic therapy: beyond drug acquisition cost. Clin Ther. 1996 Jul-Aug;18(4):716-25; discussion 702. doi: 10.1016/s0149-2918(96)80222-0. PMID 8879899
- [Background] Patel UC, McKissic EL, Kasper D, Lentino JR, Pachucki CT, Lee T, Lopansri BK. Outcomes of ceftriaxone use compared to standard of therapy in methicillin susceptible staphylococcal aureus (MSSA) bloodstream infections. Int J Clin Pharm. 2014 Dec;36(6):1282-9. doi: 10.1007/s11096-014-9999-5. Epub 2014 Sep 4. PMID 25186790
- [Background] Wieland BW, Marcantoni JR, Bommarito KM, Warren DK, Marschall J. A retrospective comparison of ceftriaxone versus oxacillin for osteoarticular infections due to methicillin-susceptible Staphylococcus aureus. Clin Infect Dis. 2012 Mar 1;54(5):585-90. doi: 10.1093/cid/cir857. Epub 2011 Dec 5. PMID 22144536
- [Background] Winans SA, Luce AM, Hasbun R. Outpatient parenteral antimicrobial therapy for the treatment of methicillin-susceptible Staphylococcus aureus: a comparison of cefazolin and ceftriaxone. Infection. 2013 Aug;41(4):769-74. doi: 10.1007/s15010-013-0477-0. Epub 2013 May 19. PMID 23686435